CLINICAL TRIAL: NCT06243523
Title: The Effect of Psychoeducation Based on Neuman's Systems Model on the Psychological Distress and Coping With Stress of the Spouses of Patients in Intensive Care Unit
Brief Title: The Effect of Psychoeducation Based on NSM on the Psychological Distress and Coping of the Spouses of Patients in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Yeliz Karaçar, Research Assistant, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-172
Record Dates: First submitted 2024-01-24; First posted 2024-02-06 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Psychological Distress; Stress, Psychological
Keywords: Neuman Systems Model; Psychoeducation; Psychological distress; Coping with stress; Intensive care unit; Stress management
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: This study is mixed methods research that combines both exploratory mixed and nested action research phases of a multi-phase mixed design. In the first phase; It is planned to develop a stress management psychoeducation program based on Neuman's Systems Model based on the literature. In the second phase; It is planned to conduct technical action research based on the radical structuralist paradigm, one of the types of action research.
  It was planned to use the criterion sampling method, one of the purposeful sampling methods, in determining the sample of the research. The psychoeducation program will be implemented in six sessions with individual interviews lasting approximately 45-60 minutes, three times a week for the spouses of patients in intensive care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Action group (Other): The action intervention of this research is the implementation of a stress management psychoeducation program based on Neuman's Systems Model for the spouses of patients hospitalized in the intensive care unit.
  Interventions: Behavioral: The stress management psychoeducation program based on Neuman's Systems Model

INTERVENTIONS:
Behavioral: The stress management psychoeducation program based on Neuman's Systems Model — The stress management psychoeducation program will be implemented in six sessions with individual interviews lasting approximately 45-60 minutes, three times a week for the spouses of patients in intensive care. The first session includes the meeting and introduction of the psychoeducation program. The second session includes the adaptation process to the intensive care unit. The third, fourth and fifth sessions include methods of coping with stress. The sixth session includes evaluation and termination of the psychoeducational program. Quantitative data of the research will be collected with the pre-action and post-action Psychological Distress Scale and the Stress Coping Styles Scale. Qualitative data of the research will be collected through semi-structured individual in-depth interviews conducted after the action.

SUMMARY:
The aim of action research this study is to examine the effect of psychoeducation based on Neuman's Systems Model on psychological distress and coping with the stress of spouses of patients in the intensive care unit. The questions of this research are listed below.

What can be done to reduce the psychological distress of spouses of patients in the intensive care unit? What can be done to increase the active coping with the stress of spouses of patients in the intensive care unit? How to structure a stress management psychoeducational program based on Neuman's Systems Theory for spouses of patients in the intensive care unit? Does a stress management psychoeducation program based on Neuman's Systems Theory reduce the psychological distress of spouses of patients in the intensive care unit? Does a stress management psychoeducational program based on Neuman's Systems Theory increase active coping with the stress of spouses of patients in intensive care?

DETAILED DESCRIPTION:
This study is mixed methods research that combines both exploratory mixed and nested action research phases of a multi-phase mixed design. In the first phase; It is planned to develop a stress management psychoeducation program based on Neuman's Systems Model based on the literature. In the second phase; It is planned to conduct technical action research based on the radical structuralist paradigm, one of the types of action research.

The study will be conducted with spouses of patients hospitalized in the Adult Intensive Care Unit of a State Hospital between January and March 2024.

It was planned to use the criterion sampling method, one of the purposeful sampling methods, in determining the sample of the research. The psychoeducation program will be implemented in six sessions with individual interviews lasting approximately 45-60 minutes, three times a week for the spouses of patients in intensive care. The first session includes the meeting and introduction of the psychoeducation program. The second session includes the adaptation process to the intensive care unit. The third, fourth and fifth sessions include methods of coping with stress. The sixth session includes evaluation and termination of the psychoeducational program.

Quantitative data of the research will be collected with the pre-action and post-action Psychological Distress Scale and the Stress Coping Styles Scale. Qualitative data of the research will be collected through semi-structured individual in-depth interviews conducted after the action. Quantitative data will be analyzed with the SPSS 25.0 package program. Continuous variables will be given as mean ± standard deviation and categorical variables will be given as number and percentage. Since non-parametric test assumptions are met in comparing the differences between psychological distress and styles of coping with stress (n<30), it will be analyzed with the Wilcoxon test. P <0.05 will be considered statistically significant. Analysis of qualitative data will be done with content analysis in Nvivo 11 qualitative data analysis program.

ELIGIBILITY:
Inclusion Criteria:

* Being the spouse of an individual with a critical illness and intubated who had an unplanned admission to the ICU for 48-72 hours or longer
* Being over 18 years of age
* Speaking Turkish

  --Not having hearing, visual, physical, or mental disabilities
* Agreeing to participate in the research verbally and in writing

Exclusion Criteria:

* Having a psychiatric illness or cognitive disorder,
* Having sensory loss related to vision, hearing, and speech,
* Being involved in another research that uses a similar method or that may affect the results of the study,
* Being included in any psychosocial support program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Kessler Psychological Distress Scale | Before action (beginning) and after action (two weeks after the beginning)
  Average score of the Kessler Psychological Distress Scale: The lowest score from the scale can be 10 and the highest score can be 50. Higher scores indicate more mental distress. Psychological distress levels according to the total score obtained from this scale; 10-19 points are interpreted as possible good, 20-24 points as possible mild mental disorder, 25-29 points as possible moderate mental disorder, and 30-50 points as possible severe mental disorder.

SECONDARY OUTCOMES:
Stress Coping Styles Scale | Before action (beginning) and after action (two weeks after the beginning)
  Average score of the Stress Coping Styles Scale: The scores obtained from the items belonging to each sub-dimension in the scale are added separately and divided by the total number of items belonging to that sub-dimension to obtain the average score for each sub-dimension. Scale Self-Confident Approach (7 items), Optimistic Approach (5 items), Helpless Approach (8 items); It consists of Submissive Approach (6 items) and Social Support Seeking (4 items) subscales.
  Self-confident approach, optimistic approach and social support seeking approach are active/effective coping methods aimed at solving the problem. Helpless approach and submissive approach are passive/ineffective ways of coping with emotions. A higher score indicates that that sub-dimension is used more.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz KARAÇAR, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruckholdt M, Tofler GH, Randall S, Buckley T. Coping by family members of critically ill hospitalised patients: An integrative review. Int J Nurs Stud. 2019 Sep;97:40-54. doi: 10.1016/j.ijnurstu.2019.04.016. Epub 2019 May 4. PMID 31132688
- [Background] Neuman B. The Neuman systems model in research and practice. Nurs Sci Q. 1996 Summer;9(2):67-70. doi: 10.1177/089431849600900207. PMID 8710312
- [Background] Fawcett J, Gigliotti E. Using conceptual models of nursing to guide nursing research: the case of the Neuman systems model. Nurs Sci Q. 2001 Oct;14(4):339-45. doi: 10.1177/089431840101400411. PMID 11873373
- [Background] Neslihan Partlak Gunusen, Ustun B, Gigliotti E. Conceptualization of burnout from the perspective of the Neuman systems model. Nurs Sci Q. 2009 Jul;22(3):200-4. doi: 10.1177/0894318409338685. PMID 19567724
- [Background] Abdul Halain A, Tang LY, Chong MC, Ibrahim NA, Abdullah KL. Psychological distress among the family members of Intensive Care Unit (ICU) patients: A scoping review. J Clin Nurs. 2022 Mar;31(5-6):497-507. doi: 10.1111/jocn.15962. Epub 2021 Jul 12. PMID 34254377